CLINICAL TRIAL: NCT05759078
Title: Effect of INtravenous FERRic Carboxymaltose Onmortality and Cardiovascular Morbidity, and Quality of Life in Iron Deficient Patients With Recent Myocardial infarCTion SUBTITLE Prevention of Cardiovascular Death, Heart Failure Events and Deterioration in Quality of Life With INtravenous FERRic Carboxymaltose in Iron Deficient Patients With Recent Myocardial Infarction
Brief Title: Effect of INtravenous FERRic Carboxymaltose Onmortality and Cardiovascular Morbidity, and Quality of Life in Iron Deficient Patients With Recent Myocardial infarCTion
Acronym: INFERRCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/ABM/01/00081
Record Dates: First submitted 2023-01-16; First posted 2023-03-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction, Acute
Keywords: Myocardial infarction; acute; iron deficiency; Infusion; ferric carboxymaltose
MeSH Terms: conditions — Myocardial Infarction; Iron Deficiencies | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Non-commercial, multicentre, randomised, double-blind, parallel group, placebo-controlled clinical trial. Eligible patients were randomly assigned (1:1) using a secure, central, interactive, web-based response system, to intervention FCM or placebo arm. Time of observation: minimum of 8 months up to a maximum of 36 months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A drip will be prepared by unblinded personnel using masked bottle, light brown lines for infusion, and administered immediately after preparation using a special curtain (screen).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): an i.v. 15-minute infusion of 20 mL Ferinject (containing 1000 mg of FCM) diluted in 50 mL of NaCl 0.9%
  Interventions: Drug: Ferinject
- Placebo (Placebo Comparator): 70 mL of i.v. NaCl 0.9% infusion
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Ferinject — The first dose of either FCM will be administered during the first visit on the day of randomisation (V1). Then, the participants will be reassessed at 4, 8, 12, 18, 24 and 30 months (visits V2, V3, V4, V5, V6, V7). If safety criteria are not fulfilled, a patient in the active study arm will receive i.v. NaCl 0.9% during the particular visit.
  Arms: Active
Drug: Sodium Chloride 0.9% Inj — The first dose of placebo will be administered during the first visit on the day of randomisation (V1). Then, the participants will be reassessed at 4, 8, 12, 18, 24 and 30 months (visits V2, V3, V4, V5, V6, V7).
  Arms: Placebo

SUMMARY:
Non-commercial, multicentre, randomised, double-blind, parallel group, placebo-controlled clinical trial. Eligible patients were randomly assigned (1:1) using a secure, central, interactive, web-based response system, to intervention FCM or placebo arm. Time of observation: minimum of 8 months up to a maximum of 36 months.

Primary Study Objective: Primary:

Evaluation of the effect of i.v. FCM treatment compared with placebo on the risk of death, the risk of heart failure events (HFE*) (number of events and time to first event), NTproBNP concentration and the change in quality of life (QoL) assessed using EQ-5D during the follow-up up to 36-months in patients with recent AMI and ID (with an implementation of a win ratio approach in a hierarchical descending order).

*HFE: unplanned hospitalization for HF (including unplanned visit at emergency department due to HF), ambulatory significant intensification of diuretic therapy (either starting i.v. loop diuretic or more than doubling oral loop diuretic dose or de novo initiation of oral loop diuretic therapy due to HF signs/symptoms).

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years;
2. Diagnosis of AMI (STEMI or NSTEMI) up to 4 weeks (28 days) before randomisation
3. Presence of iron deficiency (ID) defined as transferrin saturation TSAT<20% assessed within up to 4 weeks (28 days) before randomisation;
4. Presence of ≥3 factors (confirmed within up to 4 weeks before randomisation) (note: at least one of a-c must be present):

   1. LVEF ≤50%;
   2. NT-proBNP ≥400 pg/mL for subjects in sinus rhythm and NT-proBNP ≥800 pg/mL for subjects with atrial fibrillation;
   3. Clinical features of congestion/volume overload (including Killip class II or more) requiring i.v. loop diuretic use;
   4. Diagnosis of diabetes mellitus (also de novo diagnosis);
   5. Diagnosis of atrial fibrillation (any time in the past or de-novo diagnosis);
   6. Multivessel coronary disease (regardless of completeness of revascularisation during an index AMI);
   7. Not complete revascularisation or/and no reperfusion (during an index AMI);
   8. History of AMI (despite an index AMI);
   9. eGFR <60 mL/min/1.73m2; 1. Age ≥70 years.
5. Written informed consent

Exclusion criteria:

1. Subject temperature >38 ͦ C or any infection requiring antibiotic therapy within 48 hours prior to randomisation;
2. Severe, symptomatic valve disorder;
3. Urgent hospitalisation for whatever reasons (percutaneous/surgical procedure requiring hospitalisation within 4 weeks prior to randomisation).
4. Body weight <50 kg;
5. Haemoglobin <8 g/dL or >15,5 g/dL;
6. Serum ferritin >400 ng/mL;
7. Active gastroenteral bleeding;
8. Known hypersensitivity to any of the administered preparations;
9. Treatment with erythropoiesis stimulating factors, i.v. iron therapy or blood transfusion within 6 months prior to randomisation;
10. Subject has known active malignancy of any organ system, i.e., clinical evidence of current malignancy or not in stable remission for at least 3 years since completion of last treatment with exception of non-invasive basal cell carcinoma, squamous cell carcinoma of the skin or cervical intra-epithelial neoplasia;
11. Documented liver diseases;
12. Participation in a device or drug trial within 3 months prior to randomisation or 5 half-lives, whichever period is longer, prior to the screening visit;
13. Pregnancy or lactation;
14. Any situation that may prevent the test from being performed in accordance with the protocol, or the consent of the investigator to be given in writing, including alcohol, drugs or any other substance overuse or addiction.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause death assessed up to maximum 36-months follow-up; | up to 36 months
  Defined as: (with an implementation of a win ratio approach in a hierarchical descending order):
  1. Time to all-cause death assessed up to maximum 36-months follow-up;
  2. Number of HFE assessed up to maximum 36-months follow-up;
  3. Time to first HFE assessed up to maximum 36-months follow-up;
  4. Changes in serum NT-proBNP concentration from the start of the follow-up to the end of participation in the study assessed as the area under the curve;
  5. Changes in quality of life (QoL) measured using the EQ-5D questionnaire from the start of the follow-up to the end of participation in the study assessed as the area under the curve.
     * HFE: unplanned hospitalization for HF (including unplanned visit at emergency department due to HF), ambulatory significant intensification of diuretic therapy (either starting i.v. loop diuretic or more than doubling oral loop diuretic dose or de novo initiation of oral loop diuretic therapy due to HF signs/symptoms).
Number of HFE assessed up to maximum 36-months follow-up | up to 36 months
  Number of HFE
Time to first HFE assessed up to maximum 36-months follow-up | up to 36 months
  Time to first HFE
Changes in serum NT-proBNP concentration from the start of the follow-up to the end of participation in the study assessed as the area under the curve | up to 36 months
  Changes in serum NT-proBNP
Changes in quality of life (QoL) measured using the EQ-5D questionnaire from the start of the follow-up to the end of participation in the study assessed as the area under the curve | up to 36 months
  Changes in quality of life

SECONDARY OUTCOMES:
First unplanned HF hospitalisation or unplanned visit at emergency department due to HF or CV death during the follow-up (time-to-event model) | up to 36 months
  First unplanned HF hospitalisation or unplanned visit at emergency
All unplanned HF hospitalisations and unplanned visit at emergency department due to HF and CV death during the follow-up (recurrent event model); | up to 36 months
  All unplanned HF hospitalisations and unplanned visit at emergency
All unplanned HF hospitalisations and unplanned visit at emergency department due to HF during the follow-up (recurrent event model) | up to 36 months
  All unplanned HF hospitalisations and unplanned visit at emergency department
All unplanned HF hospitalisations during the follow-up (recurrent event model); | up to 36 months
  All unplanned HF hospitalisations
CV death during the follow-up | up to 36 months
  CV death

OTHER OUTCOMES:
First unplanned CV hospitalisation or CV death during the follow-up (time-to-event model); | up to 36 months
  First unplanned CV hospitalisation or CV death during the follow-up
All unplanned CV hospitalisations and CV death during the follow-up (recurrent event model); | up to 36 months
  All unplanned CV hospitalisations and CV death during the follow-up
All unplanned CV hospitalisations during the follow-up (recurrent event model); | up to 36 months
  All unplanned CV hospitalisations during the follow-up (recurrent event model);
Non-CV death during the follow-up | up to 36 months
  Non-CV death during the follow-up
All-cause death during the follow-up up | up to 36 months
  All-cause death during the follow-up
Ambulatory significant intensification of diuretic therapy during the follow-up | up to 36 months
  Ambulatory significant intensification of diuretic therapy (either starting i.v. loop diuretic or more than doubling oral loop diuretic dose or de novo initiation of oral loop diuretic therapy due to HF signs/symptoms) during the follow-up.
Changes in serum NT-proBNP concentration assessed as the area under the curve during the follow-up; | up to 36 months
  Changes in serum NT-proBNP concentration assessed as the area under the curve during the follow-up;
Changes in quality of life (QoL) measured using the EQ-5D questionnaire assessed as the area under the curve during the follow-up; | up to 36 months
  Changes in quality of life (QoL) measured using the EQ-5D questionnaire assessed as the area under the curve during the follow-up;
Cost-effectiveness measures during the follow-up | up to 36 months
  Cost-effectiveness measures during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ponikowski, Principal Investigator — Wroclaw Medical University
Locations (43):
- Poland (43):
  - Vitamed Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Regionalny Szpital Specjalistyczny im. dr Wł. Biegańskiego w Grudziądzu, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Wojewódzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun, Kuyavian-Pomeranian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca Małopolskie Centrum Sercowo-Naczyniowe, Chrzanów, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. SS im. Henryka Klimontowicza w Gorlicach, Gorlice, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. J. Dietla w Krakowie, Krakow, Lesser Poland Voivodeship
  - Podhalański Szpital Specjalistyczny im. Jana Pawła II w Nowym Targu, Nowy Targ, Lesser Poland Voivodeship
  - Medicome Sp. z o.o., Oświęcim, Lesser Poland Voivodeship
  - Szpital Wojewódzki im. św. Łukasza SP ZOZ w Tarnowie, Tarnów, Lesser Poland Voivodeship
  - Zespół Opieki Zdrowotnej w Kłodzku, Kłodzko, Lower Silesian Voivodeship
  - Uniwersytecki Szpital kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - 4. Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ, Wroclaw, Lower Silesian Voivodeship
  - Dolnośląski Szpital Specjalistyczny im. T. Marciniaka - Centrum Medycyny Ratunkowej, Wroclaw, Lower Silesian Voivodeship
  - Wielospecjalistyczny Szpital SP ZOZ w Zgorzelcu, Zgorzelec, Lower Silesian Voivodeship
  - 4Cardia Sp. z o.o., Kraśnik, Lublin Voivodeship
  - 1. Wojskowy Szpital Kliniczny z Polikliniką Samodzielny Publiczny Zakład Opieki Zdrowotnej w Lublinie, Lublin, Lublin Voivodeship
  - Ośrodek Kardiologii Inwazyjnej IKARDIA Sp. z o.o., Nałęczów, Lublin Voivodeship
  - Szpital Uniwersytecki imienia Karola Marcinkowskiego w Zielonej Górze Sp. z o. o., Zielona Góra, Lubusz Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Bródnowski Sp. z o.o., Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny - Państwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca Centrum Sercowo-Naczyniowe w Kędzierzynie Koźlu, Kędzierzyn-Koźle, Opole Voivodeship
  - Centrum Kardiologii w Kluczborku Scanmed S.A., Kluczbork, Opole Voivodeship
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole, Opole Voivodeship
  - Centrum Opieki Medycznej w Jarosławiu, Jarosław, Podkarpackie Voivodeship
  - Centrum Kardiologii Inwazyjnej Elektroterapii i Angiologii w Krośnie, Krosno, Podkarpackie Voivodeship
  - Uniwersyteckim Centrum Kliniczne w Gdańsku, Gdansk, Pomeranian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca Centrum Kardiologiczno-Angiologiczne w Sztumie, Sztum, Pomeranian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. Janusza Korczaka w Słupsku Sp. z o.o., Słupsk, Pomeranian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca Centrum Kardiologii i Kardiochirurgii w Bielsku-Białej, Bielsko-Biala, Silesian Voivodeship
  - Polsko-Amerykańskie Kliniki Serca, X Oddział Kardiologii Inwazyjnej, Elektrofizjologii i Elektrostymulacji w Tychach, Tychy, Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 2 PUM w Szczecinie, Szczecin, West Pomeranian Voivodeship
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewódzki Szpital Specjalistyczny w Legnicy, Legnica
  - Samodzielny Publiczny Zespół Zakładów Opieki Zdrowotnej im. dr Wojciecha Oczko w Przasnyszu, Przasnysz
  - Wojewódzki Szpital im. Św. Ojca Pio, Przemyśl
  - Szpital Specjalistyczny Ducha Świętego w Sandomierzu, Sandomierz
  - Medicover Sp z o.o., Warsaw
  - Szpital Specjalistyczny w Zabrzu Sp. z o.o., Zabrze
  - Śląskie Centrum Chorób Serca w Zabrzu, Zabrze
  - Nzoz Salusmed, Lodz, Łódź Voivodeship
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz, Łódź Voivodeship
  - Polsko-Amerykańskie Kliniki Serca Centrum Kardiologii Med-Pro, Zgierz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: INFERRCT study website — https://inferrct.umw.edu.pl/